CLINICAL TRIAL: NCT01286662
Title: In Modern Era, Recurrent Desmoids Determine Outcome in Patients With Gardner Syndrome: A Cohort Study of Three Generations of an Adenomatous Polyposis Coli (APC-) Mutation-Positive Family Across 30 Years
Brief Title: A Cohort Study of Patients Treated With Brachytherapy for Selected Desmoid Patients in Gardner Syndrome
Status: Completed | Type: Observational
Sponsor: Triemli Hospital (Other)
Responsible Party: Matthias Turina, Triemli Hospital
Other Study IDs: TriemliH
Record Dates: First submitted 2011-01-25; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Gardner Syndrome; Colorectal Carcinoma; Desmoid Tumor
Keywords: gardner syndrome; colorectal carcinoma; desmoid tumor; resection; colon
MeSH Terms: conditions — Gardner Syndrome; Colorectal Neoplasms; Desmoid Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the long-term outcome in a cohort of Gardner-Syndrome patients receiving prophylaxis and treatment for intestinal and non-intestinal tumors.

DETAILED DESCRIPTION:
Since 1978, we have been following a family of 105 descendants with Gardner Syndrome (GS). Mutation carriers were screened by endoscopy, and colorectal resection was performed upon pending malignancy. Resectable desmoid tumors were excised, whereas large tumors of the abdominal wall were treated by a combination of brachytherapy (BT) and radiotherapy (RT). Outcome was analyzed with respect to length of tumor-free survival, and morbidity from surgery or radiotherapy. Results: 37 of 105 family members have GS. Preventive colorectal resections were performed in 16 patients (15%), with one death due to subsequent gastric cancer. In 4 patients who denied screening endoscopy, invasive tumors of the colon (3 patients) and stomach (one patient each) developed. Of 33 desmoid tumors, 10 (30%) were located in the mesentery, 17 (52%) in the abdominal wall, and 6 (18%) in extra-abdominal sites. Excision of 12 desmoids was performed in 8 patients (36%), and 4 were treated by a combination of BT and RT. Following BT/RT, all patients showed full or partial remission.

ELIGIBILITY:
Inclusion Criteria:

* family with an identical adenomatous polyposis coli (APC-) germ line mutation

Exclusion Criteria:

* negative testing for adenomatous polyposis coli (APC-) germ line mutation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Since 1978, we have been following a family of 105 descendants with Gardner syndrom. APC (adenomatous polyposis coli) mutation carriers were screened by endoscopy, and colorectal resection was performed upon pending malignancy. Desmoid tumors were treated by excision or radiotherapy and brachytherapy.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 1978-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
mortality | 1978-2010 (as long as patients live)

SECONDARY OUTCOMES:
incidence of colorectal carcinoma | 1978-2010 (entire patient life)
Incidence of desmoid tumors | 1978-2010 (entire patient life)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Turina, MD PhD, Principal Investigator — Triemli Hospital; Hans P Simmen, MD, Study Director — University of Zurich Hospital

REFERENCES:
- [Derived] Turina M, Pavlik CM, Heinimann K, Behrensmeier F, Simmen HP. Recurrent desmoids determine outcome in patients with Gardner syndrome: a cohort study of three generations of an APC mutation-positive family across 30 years. Int J Colorectal Dis. 2013 Jun;28(6):865-72. doi: 10.1007/s00384-012-1600-x. Epub 2012 Nov 1. PMID 23114473